CLINICAL TRIAL: NCT00906711
Title: Analysis of Balance in the Aging Process
Status: Completed | Type: Observational
Sponsor: Universidade de Franca (Other)
Responsible Party: Lislei Jorge Patrizzi, Universidade de Franca
Other Study IDs: 0081/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Aging
Keywords: Aging; Postural Balance

STUDY DESIGN:
Biospecimen Retention: The evaluation instruments are the Berg Balance Scale (BBS), the Performance Oriented Mobility Assessment (POMA), the Unipodal Support Test, the Functional Reach Test and the Romberg's Test.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: (G1): 10 - 18 years old
- Group II: (G2): 20 - 35 years old
- Group III: (G3): 45 - 60 years old
- Group IV: (G4): 65 - 85 years old

SUMMARY:
Introduction: While growing older, it is possible to notice a decrease in the functional and physiological reserves in the organism which impairs the the abilities in the elderly in doing some tasks. A simple balance becomes a challenge.

Objective: To evaluate the functional balance in the aging process.

Methods: The group was formed by 48 people from 10 to 85 years old. The evaluation instruments are the Berg Balance Scale (BBS), the Performance Oriented Mobility Assessment (POMA), the Unipodal Support Test, the Functional Reach Test and the Romberg's Test.

DETAILED DESCRIPTION:
48 individuals of both sexes and aged between 10 and 85 years were chosen. These individuals were divided according to age, into four groups (each group containing 12 individuals, 6 men and 6 women): Group I (G1): 10 - 18, Group II (G2): 20 - 35; Group III (G3): 45 - 60, Group IV (G4): 65 - 85.

The instruments used for assessment of the balance were: (1) Berg Scale - consists of 14 items with common activities of daily life, with progressive degree of difficulty (2) Assessment of Gait and Balance for Performance Oriented (POMA), consists of a protocol that evaluates the static and dynamic balance, with operations similar to the activities of daily living, (3) Test Support Unipodal; (4) adapted Functional Reach Test, which assesses the stability in the standing position, (5) Test and Romberg Romberg's test Romberg-Barré or sensitized conducted in stable and unstable soil, and all positions were first with open eyes and then with closed eyes. The duration of each exposure was 30 seconds, with different positioning of the feet.

ELIGIBILITY:
Inclusion Criteria:

* Absence of the basic pathology that interferes directly in the balance

Exclusion Criteria:

* Neurological changes
* Cognitive impairment
* Orthopedic injury
* Use of orthoses for lower limb
* Obesity
* Exercise frequently (more than twice a week)
* The bearer of any commitment to stay in their standing position

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants were selected in dependency of Unifran (University of France) and the homes of the neighborhood. The choice of groups was based according to the degree of functionality and independence in order to analyze the lack of balance in the process of aging.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Study Director — Universidade de Franca